CLINICAL TRIAL: NCT01926145
Title: DenHeart - Self-reported Health and Quality of Life at Hospital Discharge From a Heart Centre in Denmark
Acronym: DenHeart
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: University Hospital, Gentofte, Copenhagen (Other); Odense University Hospital (Other); Aalborg University Hospital (Other); Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Selina Kikkenborg Berg, Ph.D., Rigshospitalet, Denmark
Other Study IDs: DenHeart
Record Dates: First submitted 2013-07-29; First posted 2013-08-20 (Estimated); Last update posted 2015-06-10 (Estimated); Status verified 2015-06

CONDITIONS: All Conditions Treated at the Heart Centres

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The objective of this study is to describe: 1) Differences in perceived health at hospital discharge between diagnostic groups and in-hospital predicting factors. 2) Perceived health at hospital discharge as a predictor of morbidity and mortality after 1 and 3 years. 3) The association between perceived health, sick leave and health care utilization.

The five heart centres in Denmark diagnose and treat about 50.000 patients with different diagnoses every year and offer both invasive and non-invasive treatment.

Perceived health status is measured by self-reported health, quality of life, anxiety and depression and symptoms. Knowledge about perceived health status can help to guide inpatient practise and outpatient follow-up. Furthermore, it can be used to evaluate differences between diagnostic groups, regional differences and predicting factors for perceived health status at hospital discharge and long term morbidity and mortality. Also economic analysis of healthcare utilisation and work ability status are possible.

Five Danish heart centres (Rigshospitalet, Gentofte Hospital, Odense University Hospital, Aarhus University Hospital and Aalborg University Hospital) are all including patients from April 2013 to April 2014. All patients discharged or transferred from one of the heart centres are potential participants in the study. Patients are unselected and consecutively included at hospital discharge. Included patients will be asked to complete and return a questionnaire before they leave the hospital.

The following questionnaires will be used to measure the perceived health status of the patients at hospital discharge: SF-12, Hospital Anxiety and Depression Scale, EQ-5D, Brief Illness Perception Questionnaire, HeartQoL and Edmonton Symptom Assessment Scale. Furthermore 14 ancillary about health and health behaviour are included in the questionnaire. This amounts to a total of 62 items in the questionnaire.

The DenHeart study data collection, database development and reporting of primary outcomes are funded by the five participating heart centres in Denmark. Further funding for registry data, analyses and reporting will be applied for in external funds.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized at one of the five heart centres
* Able to fill out the questionnaire

Exclusion Criteria:

* <18 years
* No Danish CPR number
* For ethical reasons unconscious patients are also excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients discharged or transferred from one of the heart centres are potential participants in the study. The diagnostic groups include ischemic heart disease, heart failure, arrhythmia, heart valve disease, endocarditis, congenital heart disease and heart transplantation.
Sampling Method: Non-Probability Sample
Enrollment: 16712 (Actual)
Dates: Start 2013-04; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Self-reported health measured by SF-12 | Baseline

SECONDARY OUTCOMES:
Hospital Anxiety and Depression Scale | Baseline
EQ-5D | Baseline
Brief Illness Perception Questionnaire | Baseline
HeartQoL | Baseline
Edmonton Symptom Assessment Scale | Baseline

OTHER OUTCOMES:
Morbidity and mortality after 1 and 3 years | 1 and 3 years after baseline
Sick leave and health care utilization | 1 and 3 years after baseline

CONTACTS AND LOCATIONS:
Overall Officials: Selina K Berg, Ph.D., Principal Investigator — Rigshospitalet, Denmark
Locations (5):
- Denmark (5):
  - Aalborg University Hospital, Aalborg
  - Aarhus University Hospital, Aarhus
  - Gentofte Hospital, Copenhagen
  - Rigshospitalet, Copenhagen University Hospital, Copenhagen
  - Odense University Hospital, Odense

REFERENCES:
- [Derived] Wagner MK, Christensen AV, Hassager C, Stenbaek DS, Ekholm O, Borregaard B, Thrysoee L, Rasmussen TB, Thorup CB, Mols RE, Juel K, Berg SK. Sex Differences in Patient-Reported Outcomes in the Immediate Recovery Period After Resuscitation: Findings From the Cross-sectional DenHeart Survey. J Cardiovasc Nurs. 2023 May-Jun 01;38(3):279-287. doi: 10.1097/JCN.0000000000000914. Epub 2022 Apr 27. PMID 37027133
- [Derived] Dalsgaard JL, Hansen MS, Thrysoee L, Ekholm O, Thorup CB, Mols RE, Rasmussen TB, Christensen AV, Berg SK, Pedersen AK, Jensen LO, Mogensen CB, Borregaard B. Self-reported health and adverse outcomes among women living with symptoms of angina or unspecific chest pain but no diagnosis of obstructive coronary artery disease-findings from the DenHeart study. Eur J Cardiovasc Nurs. 2023 Jul 19;22(5):506-515. doi: 10.1093/eurjcn/zvac085. PMID 36124692
- [Derived] Mols RE, Borregaard B, Logstrup BB, Rasmussen TB, Thrysoee L, Thorup CB, Christensen AV, Ekholm O, Rasmussen AA, Eiskjaer H, Risor BW, Berg SK. Patient-reported outcome is associated with health care costs in patients with ischaemic heart disease and arrhythmia. Eur J Cardiovasc Nurs. 2023 Jan 12;22(1):23-32. doi: 10.1093/eurjcn/zvac030. PMID 35543021
- [Derived] Risom SS, Thygesen LC, Rasmussen TB, Borregaard B, Norgaard MW, Mols R, Christensen AV, Thorup CB, Thrysoee L, Juel K, Ekholm O, Berg SK. Association Between Risk Factors and Readmission for Patients With Atrial Fibrillation Treated With Catheter Ablation: Results From the Nationwide DenHeart Study. J Cardiovasc Nurs. 2023 Jan-Feb 01;38(1):E31-E39. doi: 10.1097/JCN.0000000000000900. Epub 2022 Mar 10. PMID 35275884
- [Derived] Christensen AV, Cromhout PF, Jorgensen MB, Ekholm O, Juel K, Svendsen JH, Rasmussen TB, Borregaard B, Mols RE, Thrysoee L, Thorup CB, Berg SK. Cause of Death Among Cardiac Patients With and Without Anxiety. J Cardiovasc Nurs. 2022 Sep-Oct 01;37(5):E122-E128. doi: 10.1097/JCN.0000000000000832. PMID 34224466
- [Derived] Nielsen SN, Rasmussen TB, Lassen JF, Berg SK, Thrysoee L, Moller JE, Jensen LO, Thuesen AL, Christensen AV, Ekholm O, Mols R, Thorup CB, Borregaard B. The association between self-reported health status and adverse events: a comparison among coronary artery bypass grafting (CABG) versus percutaneous coronary intervention (PCI). Qual Life Res. 2020 Nov;29(11):3017-3029. doi: 10.1007/s11136-020-02573-8. Epub 2020 Aug 28. PMID 32857268
- [Derived] Christensen AV, Dixon JK, Juel K, Ekholm O, Rasmussen TB, Borregaard B, Mols RE, Thrysoe L, Thorup CB, Berg SK. Psychometric properties of the Danish Hospital Anxiety and Depression Scale in patients with cardiac disease: results from the DenHeart survey. Health Qual Life Outcomes. 2020 Jan 7;18(1):9. doi: 10.1186/s12955-019-1264-0. PMID 31910859
- [Derived] Berg SK, Svanholm J, Lauberg A, Borregaard B, Herning M, Mygind A, Christensen AV, Christensen AI, Ekholm O, Juel K, Thrysoe L. Patient-reported outcomes at hospital discharge from Heart Centres, a national cross-sectional survey with a register-based follow-up: the DenHeart study protocol. BMJ Open. 2014 May 2;4(5):e004709. doi: 10.1136/bmjopen-2013-004709. PMID 24793253